CLINICAL TRIAL: NCT01940068
Title: A Double-blind Randomized Controlled Trial of a Thickened Amino-acid-based Formula in Children Allergic to Cow's Milk and to Protein Hydrolysates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-UP05-E1
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Cow Milk Allergy
Keywords: Hypersensitivity; Milk Hypersensitivity; Immune System Diseases; Food Hypersensitivity
MeSH Terms: conditions — Milk Hypersensitivity; Hypersensitivity; Immune System Diseases; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Thickened Amino acid based formula (Experimental)
  Interventions: Dietary Supplement: Amino acid based formula
- Amino acid based formula (Active Comparator)
  Interventions: Dietary Supplement: Amino acid based formula

INTERVENTIONS:
Dietary Supplement: Amino acid based formula

SUMMARY:
The purpose of this study is to evaluate the impact of a new Amino-acid based formula on allergic symptoms and growth of infants with cow's milk protein allergy and intolerant to extensively hydrolysed formulas;

ELIGIBILITY:
Inclusion Criteria:

* less than 18 months old
* with a proven cow's milk protein allergy by a double blind placebo controlled food challenge or a positive Skin prick test (>=6mm) or specific immunoglobulin E >= 5 kilo-unit/L or combination
* still symptomatic while fed an extensively hydrolysed formula

Exclusion Criteria:

* Exclusively breast fed infants
* non allergic digestive enteropathy

Ages: 2 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of withdrawal for intolerance | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Necker Children's Hospital, Paris, France

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765
- [Derived] Dupont C, Kalach N, Soulaines P, Bradatan E, Lachaux A, Payot F, De Blay F, Guenard-Bilbault L, Hatahet R, Mulier S, Kapel N, Waligora-Dupriet AJ, Butel MJ. Safety of a New Amino Acid Formula in Infants Allergic to Cow's Milk and Intolerant to Hydrolysates. J Pediatr Gastroenterol Nutr. 2015 Oct;61(4):456-63. doi: 10.1097/MPG.0000000000000803. PMID 25844709
- [Derived] Dupont C, Kalach N, Soulaines P, Bradatan E, Lachaux A, Payot F, de Blay F, Guenard-Bilbault L, Hatahet R, Mulier S. A thickened amino-acid formula in infants with cow's milk allergy failing to respond to protein hydrolysate formulas: a randomized double-blind trial. Paediatr Drugs. 2014 Dec;16(6):513-22. doi: 10.1007/s40272-014-0097-x. PMID 25446768